CLINICAL TRIAL: NCT01153997
Title: A Randomised, Placebo-controlled Single-dose, Parallel-group, Double-blind Trial Evaluating Safety and Pharmacokinetics of Recombinant Factor XIII in Healthy Japanese Subjects
Brief Title: Safety of Recombinant Factor XIII (rFXIII) in Healthy Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1810-3733; U1111-1114-8989 (Other: WHO); 101192 (Registry Identifier: JAPIC)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Acquired Bleeding Disorder; Cardiac Surgery Requiring Cardiopulmonary Bypass; Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental)
  Interventions: Drug: catridecacog
- B (Experimental)
  Interventions: Drug: catridecacog
- C (Placebo Comparator)
  Interventions: Drug: placebo
- D (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: catridecacog — Single rFXIII dose (12 IU/kg). Administered via slow intravenous (i.v.) push at a rate not exceeding two mL per minute.
  Arms: A
Drug: placebo — Single rFXIII placebo dose (12 IU/kg). Administered via slow intravenous (i.v.) push at a rate not exceeding two mL per minute.
  Arms: C
Drug: catridecacog — Single rFXIII dose (35 IU/kg). Administered via slow intravenous (i.v.) push at a rate not exceeding two mL per minute.
  Arms: B
Drug: placebo — Single rFXIII placebo dose (35 IU/kg). Administered via slow intravenous (i.v.) push at a rate not exceeding two mL per minute.
  Arms: D

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to investigate the safety profile of recombinant factor XIII (rFXIII) assessed by the occurrence of adverse events in healthy Japanese subjects. In addition pharmacokinetic parameters will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Good general health based on assessment of medical history, physical examination, ECG (electrocardiogram) and clinical laboratory data at screening, as judged by the physician
* Body mass index (BMI) between 18.0-27.0 kg/m2 (both inclusive)

Exclusion Criteria:

* The receipt of any investigational products for coagulation factor protein within 6 months prior to trial start (screening)
* Known or suspected allergy to yeast
* Known bleeding or hematologic disorder
* Significant history of alcoholism or drug/chemical abuse as judged by the physician or positive result in the alcohol breath test/screen of drugs at the trial start (screening)
* Smoking more than 10 cigarettes/day or equivalent
* Not able or willing to refrain from smoking whenever required for the trial procedures
* Habitual excessive consumption of methylxanthine-containing beverages and foods (coffee, tea, soft drinks such as cola, chocolate) as judged by the physician
* Excessive consumption of a diet deviating from a normal diet as judged by the physician
* Strenuous exercise as judged by the physician within 4 days prior to trial start (screening)
* Surgery or trauma with significant blood loss (500 mL or more blood) within 3 months prior to trial start (screening)
* Males who are sexually active and not surgically sterilised, who or whose partner are not using adequate contraceptive methods. Adequate contraceptive measures include that the subject uses a condom during intercourse or that the partner practices adequate conception (sterilisation, hormonal intrauterine devices and oral contraceptives).

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of serious adverse events | from first trial related activity (visit 1) and up to 28 days (visit 8) after dosing
Occurrence of non-serious adverse events | from first trial related activity (visit 1) and up to 28 days (visit 8) after dosing

SECONDARY OUTCOMES:
AUC (area under the curve) from time zero to 28 days | at day 28

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Fukuoka, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com